CLINICAL TRIAL: NCT00082043
Title: The Effects of Dutasteride on Mood, HPA Axis, and Serum Allopregnanolone Levels in Women With Menstrual-Related Mood Disorders and Controls
Brief Title: Dutasteride to Treat Women With Menstrually Related Mood Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 040139; 04-M-0139
Record Dates: First submitted 2004-04-28; First posted 2004-04-28 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-02-05

CONDITIONS: Premenstrual Syndrome; PMS; Healthy; Depression
Keywords: Neurosteroids; 5 Alpha-Reductase Inhibitor; Depression; Menstrual Cycle; Gonadal Steroids; Menstrual Cycle Related Mood Disorder; MRMD; Healthy Volunteer
MeSH Terms: conditions — Premenstrual Syndrome; Depression | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Dutasteride 2.5 mg by mouth daily for one month
  Interventions: Drug: Dutasteride
- 2 (Placebo Comparator): Placebo oral capsule for two months
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Dutasteride
  Arms: 1
Drug: Placebo oral capsule
  Arms: 2

SUMMARY:
This study will explore the effects of dutasteride on mood and the stress response across the menstrual cycle. Dutasteride blocks production of neurosteroids-hormones that help regulate the stress response systems. These systems may be disturbed in women with menstrually related mood disorders (MRMD). The effects of the drug will be compared in women with and without MRMD to determine how neurosteroids regulate mood and the stress response across the menstrual cycle. Dutasteride is approved by the Food and Drug Administration to treat benign prostatic hyperplasia (excess growth of the prostate gland) in men.

Menstruating women 30 to 45 years of age with and without MRMD may be eligible for this study. Candidates are screened with a medical and psychiatric history, physical examination, screening for symptoms of depression, and routine blood and urine tests. Participants are required to use barrier contraception (condoms or diaphragm) during the 3-month study and 6-month follow-up.

Participants undergo the following tests and procedures:

* Dutasteride or placebo treatment: Participants receive 1 month of dutasteride and 2 months of placebo. Neither the participants nor the investigators know when the subject is taking the active medication or the placebo.
* Biweekly follow-up visits: Every 2 weeks during the 3-month treatment period, patients come to the NIH Clinical Center to have blood drawn and to complete mood symptoms ratings.
* Monthly follow-up visits: Participants return to the Clinical Center once a month for 6 months after the end of the treatment period to monitor hormone levels and pregnancy status.

DETAILED DESCRIPTION:
Studies of premenstrual syndrome (PMS) to date have demonstrated that the syndrome represents an abnormal response to normal physiological events. Specifically patients with PMS experience a dysphoric mood state in response to normal luteal phase levels of progesterone and additionally fail to demonstrate the augmentation of the hypothalamic-pituitary-adrenal (HPA) axis normally seen in the luteal phase. A parsimonious explanation for the dysregulation of both mood and HPA axis function in PMS is that both are mediated by abnormal levels of or response to the progesterone neurosteriod metabolite, allopregnanolone. Both exposure to and withdrawal from allopregnanolone have been shown to precipitate adverse mood states in animal studies, presumably consequent to induced conformational changes in the GABA(A) receptor (increased alpha-4 subunit) that impair GABA receptor function. This impairment of GABA receptor function may also be associated with loss of restraint of HPA axis activity and hence may underlie the luteal phase increases in HPA activity in normal women. In this protocol, we propose to block conversion of progesterone to allopregnanolone in women with menstrual-related mood disorder (MRMD; equivalent in most reports to a severe form of PMS called premenstrual dysphoric disorder (PMDD)) and in normal (control) women. We will block progesterone metabolism (and hence exposure to allopregnanolone) with a newly approved 5 alpha-reductase inhibitor, dutasteride. We hypothesize the following: 1) Elimination of exposure to allopregnanolone in women with MRMD will eliminate dysphoric mood in the luteal phase; 2) Elimination of exposure of normal control women to allopregnanolone will eliminate the luteal phase enhancement of stimulated stress axis activity response.

These hypotheses, if confirmed, will increase the precision with which we can dissect the pathophysiological mechanisms involved in MRMD and in menstrual-related stress physiology.

In this protocol, our study objectives are as follows: Primary Objectives: 1) Determine whether suppression of neurosteroid synthesis will diminish mood symptoms in women with MRMD. 2) Determine if suppression of neurosteroid synthesis will eliminate luteal phase-related increases in stimulated HPA axis activity in control women. Secondary Objectives: 1) Determine whether differences in response to allopregnanolone account for the divergent effects of menstrual cycle phase on HPA axis activity in patients with MRMD and controls. 2) Determine if the Dex-CRH test, like the graded stressor treadmill test, can reveal the effects of menstrual cycle phase on HPA axis function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy controls and women who meet the criteria for MRMD.

The criteria for MRMD, from Protocol 81-M-126, "The Phenomenology and Biophysiology of Menstrually Regulated Mood and Behavior Disorders," briefly are as follows:

1. History within the last two years of at least six months with menstrually-related mood or behavioral disturbances of a severity sufficient to cause at least moderate subjective distress;
2. Symptoms should have a sudden onset and offset, with symptoms most severe during the week prior to menstruation and tending to disappear abruptly on or about the first day menstruation;
3. Age 30-50 years;
4. In good physical health;
5. To qualify for study inclusion, women with MRMD will have prospectively demonstrated in at least two of three menstrual cycles a 30% worsening of mean negative mood symptoms in the premenstrual period compared to the week following menses, corrected for the range of the scales employed.

Healthy controls will have no symptoms of MRMD (confirmed prospectively), be between the ages of 30 and 50, and be in good physical health.

In addition all subjects will have a normal clinical breast exam prior to study entry.

EXCLUSION CRITERIA:

Subjects will be excluded from the study for the following reasons:

1. Pregnancy or any intent to become pregnant;
2. Medical illness, in particular diabetes, cardiac or renal disease;
3. Use of psychotropic or hormonal medications within three months prior to the study;
4. Current prescription medication use;
5. History of or current alcohol or drug abuse or dependence;
6. A history of (within the past two years) or current psychiatric disorder determined by administration of the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID);
7. Male gender;
8. Age less than 30 years; and
9. Women with a history of carcinoma of the breast, or women with a family history of the following: premenopausal breast cancer or bilateral breast cancer in a first degree relative; multiple family members (greater than three relatives) with a history of postmenopausal breast cancer.

In addition to the above, due to the long half life of dutasteride and its teratogenic effects on male fetuses, only women who have already decided to discontinue child-bearing and are willing to continue barrier contraception for 6 months after the study will be included in the protocol.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2004-03-31; Primary Completion 2014-03-06 (Actual); Study Completion 2014-03-06 (Actual)

PRIMARY OUTCOMES:
Rating Scale for Premenstrual Tension (PMTS); Daily symptom rating form (DRF); Visual Analogue Symptom (VAS) self-rating form. | Every 2 weeks for the PMTS; daily for the others.

SECONDARY OUTCOMES:
Neuroendocrine response to DEX/crh test; Beck Depression Inventory (BDI) | DEX/crf 2x second mth of tx, 1x during luteal ph & 1x during follicular ph.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E Martinez, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Halbreich U, Borenstein J, Pearlstein T, Kahn LS. The prevalence, impairment, impact, and burden of premenstrual dysphoric disorder (PMS/PMDD). Psychoneuroendocrinology. 2003 Aug;28 Suppl 3:1-23. doi: 10.1016/s0306-4530(03)00098-2. PMID 12892987
- [Background] Wittchen H -U, Becker E, Lieb R, Krause P. Prevalence, incidence and stability of premenstrual dysphoric disorder in the community. Psychol Med. 2002 Jan;32(1):119-32. doi: 10.1017/s0033291701004925. PMID 11883723
- [Background] Rubinow DR, Roy-Byrne P. Premenstrual syndromes: overview from a methodologic perspective. Am J Psychiatry. 1984 Feb;141(2):163-72. doi: 10.1176/ajp.141.2.163. PMID 6362441